CLINICAL TRIAL: NCT05859243
Title: Effects of Traditional Concurrent Training and Concurrent Training Composed by Strenght Traning and Dance Classes in Functional Performance, Cognitive Function and Quality of Life of Older Adults: a Randomized Controlled Clinical Trial
Brief Title: Effects of Two Types of Concurrent Training in Functional Performance and Cognitive Function of Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eduardo Lusa Cadore (Other)
Responsible Party: Sponsor-Investigator, Eduardo Lusa Cadore, Professor, Federal University of Rio Grande do Sul
Organization: Federal University of Rio Grande do Sul (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: uRioGrandeLAPEx
Record Dates: First submitted 2023-04-24; First posted 2023-05-15 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Aging
Keywords: Aging; Functional capacity; Physical activities
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Traditional concurrent training (Experimental): The subjects will perform two concurrent training sessions, of approximately one hour per week. Composed of strength exercises and aerobic exercise (walking outdoors and/or treadmill).
  Interventions: Behavioral: Traditional concurrent training
- Concurrent training consisting of strength training combined with dance classes (Experimental): The subjects will perform two concurrent training sessions associated with dance classes, of approximately one hour per week. Composed of strength exercises and dance classes.
  Interventions: Behavioral: Concurrent training consisting of strength training combined with dance classes
- Control (No Intervention): Subjects will be instructed to maintain their usual routine during the study period.

INTERVENTIONS:
Behavioral: Traditional concurrent training — The subjects will perform two sessions per week of traditional concurrent training, consisting of strength training followed by aerobic exercise over 12 weeks, with progressive intensities and training volumes. Each traditional concurrent training session will consist of specific warm-up performed on equipment for upper and lower limbs with a load of less than 30% of the training load. Then the bench press, low row, leg press, extension and knee flexion exercises will be performed. Participants will be instructed to perform the concentric phase of the movement in one second and the eccentric phase in two seconds. After strength training, aerobic training (walking outdoors or on a treadmill) will be performed with intensity based on the adapted BORG effort perception scale (ranged to 0 = minimum effort, to 10 = maximal effort).
  Arms: Traditional concurrent training
Behavioral: Concurrent training consisting of strength training combined with dance classes — Each concurrent training session associated with dance classes will consist of the same strength training as the traditional concurrent training group, but the traditional aerobic training will be replaced by a dance class. Each dance class will consist of a 5-minute general warm-up with joint mobility exercises and dynamic stretching. Then the main part will be performed with the elaboration of choreography, lasting approximately 20 minutes. Finally, there will be a 5-minute cool-down with stretching exercises. Classes will be held in four different dance modalities, divided into four modules.
  Arms: Concurrent training consisting of strength training combined with dance classes

SUMMARY:
The goal of this randomized controlled clinical trial is to identify and compare the impacts of traditional concurrent training and concurrent training consisting of strength training combined with dance classes on functional performance, cognitive function and quality of life in older people. The main question it aims to answer are:

• The concurrent training consisting of strength training combined with dance classes can provide similar benefits to traditional concurrent training in neuromuscular and cardiorrespiratory performance, cognitive function and quality of life in older people?

Participants will training one of the two types of concurrent training (traditional concurrent training or concurrent training consisting of strength training combined with dance classes), two times a week, over 12 weeks.

Researchers will compare traditional concurrent training, concurrent training consisting of strength training combined with dance classes and a control group without exercise to see if this modalitys of physical exercise can provide increases in neuromuscular and cardiorrespiratory performance, cognitive function and quality of life in older people.

ELIGIBILITY:
Inclusion criteria:

* Be male or female aged between 65 and 75 years old
* Do not practice regular physical exercises for at least three months
* No history of competitive sports throughout life
* Not having musculoskeletal and neurological diseases or disorders that may influence the performance of the exercises or affect the test results
* Not having health conditions in which physical exercise is contraindicated
* Achieve a score of no less than 24 on the Mini Mental State Exam
* Achieve a score of up to 9.11 on the Baecke Physical Activity Questionnaire.

Exclusion criteria:

* Miss more than 20% of training sessions
* Miss more than three workouts in a row
* Failure to attend any of the evaluations will be excluded from the study.

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 44 (Actual)
Dates: Start 2023-05-22 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Change in Dynamic balance | Baseline, 8 and 12 weeks
  Assessed by Timed Up and Go Test
Change in Cognitive function | Baseline, 8 and 12 weeks
  Assessed by Mini Exam of Mental State
Change in Self reported quality of life | Baseline, 8 and 12 weeks
  Assessed by World Health Organization Quality of Life Questionary, on a scale ranging from 26 to 130. Higher scores are considered better.
Change in Static Balance | Baseline, 8 and 12 weeks
  Assessed by One leg Stance Test
Change in Seat to Stand Capacity | Baseline, 8 and 12 weeks
  Assessed by 30s Seat to Stand Test
Change in Stairs Climb Capacity | Baseline, 8 and 12 weeks
  Assessed by 10 step climb test
Change in Leg Strenght | Baseline, 8 and 12 weeks
  Assessed by One repetition maximum knee extension test
Change in Leg Power | Baseline, 8 and 12 weeks
  Assessd by 30% and 70% of One repetition maximum knee extension Test
Change in Hand Grip Strenght | Baseline, 8 and 12 weeks
  Assessed by Hand Grip Test with Hydraulic Dynamometer
Change in Cardiorrespiratory Capacity | Baseline, 8 and 12 weeks
  Assessed by the 6 minutes walk test

SECONDARY OUTCOMES:
Change in Quadriceps muscle thickness | Baseline and 12 weeks
  Assessed by ultrasound
Change in Affectivity with the intervention | 8 and 12 weeks
  Assessed by Scale (+5 = very good, -5 = very bad)
Change in Lipid profile | Baseline and 12 weeks
  plasma concentrations of total cholesterol, HDL and triglycerides will be determined by the colorimetric method with specific kits in an automatic analyzer (Cobas C111, Roche Diagnostics, Basel, Switzerland).
Change in Specific tension of quadriceps | Baseline and 12 weeks
  Calculated by the formula: maximum knee extension strength/quadriceps muscle thickness
Change in depressive symptoms | Baseline and 12 weeks
  Measured using the Geriatric Depression Scale, that consists of 15 questions with binary answers (yes/no) and easy to understand. It ranges from zero (absence of depressive symptoms) to fifteen points (maximum score of depressive symptoms).

CONTACTS AND LOCATIONS:
Locations (1):
- Escola de Educação Física, Fisioterapia e Dança - UFRGS, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-01-30): https://cdn.clinicaltrials.gov/large-docs/43/NCT05859243/Prot_SAP_000.pdf
  • Informed Consent Form (2023-01-30): https://cdn.clinicaltrials.gov/large-docs/43/NCT05859243/ICF_001.pdf